CLINICAL TRIAL: NCT03787277
Title: CT Evaluation of Intimal Flap Mobility as a Potential Predictor of Residual Type B Dissection Evolution
Brief Title: CT Evaluation of Intimal Flap Mobility
Acronym: CT-MOBILITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7310
Record Dates: First submitted 2018-12-13; First posted 2018-12-26 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-12

CONDITIONS: Aortic Dissection Type A
Keywords: Aortic Dissection Type A; Post operative residual aortic dissection; Aneurysmal progression of the dissected aorta; Intimal flap mobility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type A aortic dissection is an emergency condition, defined by the appearance of an intimal flap within the ascending aorta. Urgent treatment is required, with surgical replacement of - at minima - the tubular portion of the ascending aorta.

After surgery, a majority of patients will still have a residual aortic dissection involving the aortic arch and/or the descending aorta. Long-term survival in these patients can be hindered by the apparition of an aneurysmal progression of the dissected aorta, with risk of rupture, thrombose and/or embolism. Consequently, this condition requires frequent follow-up imaging examinations, usually by Computed Tomography Angiography (CTA), to monitor the extension of the dissection and the diameters of the dissected aorta. Patient management is therefore based on passive follow-up of the disease, as no definitive clinical or imaging features can predict the potential evolution (or the absence of) towards an aneurysmal evolution.

Therefore, one can understand the important need for accurate predictors of aneurysmal dilatation of post-operative residual dissection.

CTA has the ability to visualize the intimal flap motion, by averaging at least 3 or 4 cardiac cycles over a non-gated arterial acquisition.

This intimal flap mobility varies greatly between patients, between the localization and the extension of the dissection, and between acute and chronic dissections. It is thought that chronic dissections with immobile flap might be less prone to aneurysmal evolution.

The investigators hypothesize that this mobility could be a prognostic marker for the evolution towards aortic dilatation: flap that would remain highly mobile after initial surgery could be an additional marker towards an aneurysmal evolution, while immobile flap could be on the contrary a marker of stability.

Intimal flap motion can already be qualitatively and quantitatively assessed in CTA when ECG-synchronization is used. However, this technique has a limited availability and significantly increases the total radiation dose, therefore limiting its use in routine practice. Being able to quantify this marker using routine non ECG-gated CTA could be a significant addition to the literature, as it is currently unknown if this is feasible/relevant.

ELIGIBILITY:
Inclusion criteria:

* Major patient (≥18 years old)
* Ascending aorta replacement for aortic dissection, between 2010 and 2015 (timeframe established to allow for a significant follow-up period after surgery)
* Residual type B dissection after surgery availability of thin-slices good quality CT angiography before (at least one) and after (at least two) the surgery.

Exclusion criteria:

* Patient expressing opposition to participating in the study
* Patient under the protection of justice
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient having ascending aorta replacement for aortic dissection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the mobility of the intimal flap with CT angiography without the use of ECG synchronization | The period from January 1st, 2010 to December 31, 2015 will be examined
  The study concerns patients operated at Strasbourg University Hospitals for the replacement of the ascending aorta for aortic dissection from 2010 to 2015

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie B - NHC, Strasbourg, France